CLINICAL TRIAL: NCT05189977
Title: A Phase 1, Open-label, Fixed-sequence, Cross-over Trial to Assess the Effects of a Single Dose of Prazosin or Propranolol in the Presence of Brexpiprazole/Sertraline at Steady-state on Blood Pressure
Brief Title: A Trial to Assess the Effects of Prazosin or Propranolol on Blood Pressure in the Presence of Brexpiprazole/Sertraline
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision to terminate the trial early was not based on safety concerns. The trial was terminated early due to some implausible blood pressure values being captured, which was the primary endpoint of the study.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 331-201-00246
Record Dates: First submitted 2021-10-22; First posted 2022-01-13 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Post-traumatic Stress Disorder (PTSD)
Keywords: Major Depressive Disorder (MDD); Post-traumatic stress disorder (PTSD); Generalized Anxiety Disorder (GAD); Panic Disorder; Social Anxiety Disorder (SAD); Obsessive-Compulsive Disorder (OCD); Mental disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major; Generalized Anxiety Disorder; Panic Disorder; Phobia, Social; Obsessive-Compulsive Disorder; Mental Disorders | interventions — Propranolol; Prazosin

STUDY DESIGN:
Intervention Model Description: • Cross-over: participants receive one of two alternative interventions during the initial phase of the study and receive the other intervention during the second phase of the study
Masking Description: • Open: no masking is used. All involved know the identity of the intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sertraline alone at steady state (Active Comparator): To assess the hemodynamic changes associated with the effects of a single dose of prazosin or propranolol in the presence of brexpiprazole + sertraline at steady state compared with a single dose of prazosin or propranolol in the presence of sertraline alone at steady state.
  Interventions: Drug: Propranolol; Drug: Prazosin
- Sertraline + brexpiprazole at steady state (Active Comparator): To assess the hemodynamic changes associated with the effects of a single dose of prazosin or propranolol in the presence of brexpiprazole + sertraline at steady state compared with a single dose of prazosin or propranolol in the presence of sertraline alone at steady state.
  Interventions: Drug: Propranolol; Drug: Prazosin

INTERVENTIONS:
Drug: Propranolol — Propranolol (tablet, oral ): 40 mg QD Day 3 and Day 21
  Intervention 1 is a single dose of prazosin administered in the presence of sertraline alone at steady state or in the presence of sertraline + brexpiprazole at steady state.
Drug: Prazosin — Prazosin (tablet, oral): 1 mg QD Day 2 and Day 20
  Intervention 2 is a single dose of propranolol administered in the presence of sertraline alone at steady state or in the presence of sertraline + brexpiprazole at steady state.

SUMMARY:
A Trial to Assess the Effects of Prazosin or Propranolol on Blood Pressure in the Presence of Brexpiprazole/Sertraline

ELIGIBILITY:
Inclusion Criteria:

* Primary Diagnostic and Statistical Manual of Mental Disorders (DSM), Fifth Edition criteria Diagnosis of Major Depressive Disorder, post-traumatic stress disorder, generalized anxiety disorder, panic disorder, social anxiety disorder or obsessive-compulsive disorder
* Must be able to receive a sertraline dose of 150 mg/day by the second screening visit (Day -15)

Exclusion Criteria

* Sexually active males or females, who could become pregnant, not agreeing to practice 2 different methods of birth control or remain abstinent during the trial and for 30 days at the end of the study
* Diagnosed hypertension (including treated or untreated hypertension), or orthostatic hypotension
* Epilepsy or a history of seizures
* History of neuroleptic malignant syndrome or serotonin syndrome.
* Primary DSM-5 diagnosis of Schizophrenia spectrum and other psychotic disorders, Bipolar and related disorders, Feeding and eating disorders (including anorexia nervosa or bulimia), Neurocognitive disorders (including but not limited to delirium, major or mild neurocognitive disorder due to Alzheimer's, Parkinson's, or traumatic brain injury)
* A significant risk of committing violent acts, serious self-harm, or suicide
* History of diabetes mellitus (type 1 or type 2)
* Subjects with any previous exposure to brexpiprazole, or subjects with chronic use of prazosin or propranolol in the 90 days prior to the screening visit or any use in the 21 days (3 weeks) prior to the screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Changes between the control and treatment periods on Day 19 vs. Day 1, Day 20 vs. Day 2, and Day 21 vs. Day 3, with prazosin or propanolol in the presence of brexpiprazole + sertraline or sertraline alone at steady state | 21 days
  Mean difference in baseline-adjusted change in systolic blood pressure (ΔΔSBP), measured in mmHg, from supine to standing positions will be assessed.
Maximum change in SBP, measured in mmHg, from supine to standing position in the presence of brexpiprazole + sertraline or sertraline alone at steady state will be assessed. | 21 days
Maximum change in diastolic blood pressure (DBP), measured in mmHg, from supine to standing position in the presence of brexpiprazole + sertraline or sertraline alone at steady state will be assessed. | 21 days
Maximum change in resting heart rate (HR), measured in beats per minute (bpm), from supine to standing position will be assessed in the presence of brexpiprazole + sertraline or sertraline alone at steady state will be assessed. | 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding sites (California, Texas, New Jersey, Minnesota), Princeton, New Jersey, United States